CLINICAL TRIAL: NCT02115724
Title: Effect of Low Childhood Socioeconomic Status (SES) on Adult Endothelial Function and Nitric Oxide Bioavailability in Vivo and ex Vivo
Brief Title: Nitric Oxide Bioavailability and Early Life Stress (NO-Stress)
Acronym: NO-Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Harris, Assistant Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NO-Stress Pro00001887; 5P01HL069999 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-16 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Disease
Keywords: Low childhood SES; Early Life Stress; Endothelial function; Flow mediated dilation; Cardiovascular disease; Subcutaneous adipose arterioles
MeSH Terms: conditions — Cardiovascular Diseases; Stress, Psychological | interventions — Ascorbic Acid; Vitamin E; Thioctic Acid; Biopsy; Nonsense Mediated mRNA Decay

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidant Cocktail (Experimental): Following an overnight fast, blood samples, flow-mediated dilation, and nitroglycerin mediated dilation (NMD; 0.4mg sub-lingual nitroglycerin spray) will be performed at baseline and 2 hours following either a single dose oral antioxidant cocktail (1000 mg Vitamin C, 600 IU vitamin E, 600 mg Alpha Lipoic Acid) or placebo on two days separated by at least 72 hours.
  Interventions: Dietary Supplement: Antioxidant cocktail; Other: Placebo; Drug: NMD; 0.4mg sub-lingual nitroglycerin spray
- Biopsy (Other): Following an overnight fast, a subcutaneous gluteal/hip fat biopsy sample will be obtained from each subject under local anesthesia, with adipose tissue (~2x1.5x1.5cm) to be harvested and placed immediately in physiological saline solution (PSS): Small arteries, 100 to 150 um in diameter, will be dissected from the fat under a dissecting microscope, transferred to an arteriographic bath chamber, and cannulated for pressurized myography.
  Interventions: Other: Biopsy

INTERVENTIONS:
Dietary Supplement: Antioxidant cocktail — Flow-Mediated Dilation will be determined at baseline and 2 hours following acute antioxidant treatment
  Other Names: Vitamin C; Vitamin E; Alpha Lipoic Acid
  Arms: Antioxidant Cocktail
Other: Biopsy — Under sterile conditions, a small incision (¼ - ½ inch) by the study doctor will be made and the piece of fat will be taken out. Fat tissue was chosen for this study because it is a big source of small blood vessels which we are studying
  Arms: Biopsy
Other: Placebo — Flow-Mediated Dilation will be determined at baseline and 2 hours following acute antioxidant treatment
  Arms: Antioxidant Cocktail
Drug: NMD; 0.4mg sub-lingual nitroglycerin spray — Nitroglycerin mediated dilation will be measured immediately following an administered 0.4mg dose of nitroglycerin spray, sub-lingual.
  Other Names: Generic name: Nitrolingual; Manufacturer: Arbor Pharmaceuticals
  Arms: Antioxidant Cocktail

SUMMARY:
Cardiovascular disease is the leading cause of death in the United States. Other studies have shown that stress, early in life, could be a risk factor for cardiovascular disease, later in life. This study will look at the effect of early life stressors on your cardiovascular health.

DETAILED DESCRIPTION:
This study will have two parts involved to investigate the role that childhood SES status has on cardiovascular health.

Part one: Subjects will give a blood sample which will be processed and analyzed. Flow mediated dilation (FMD) and Pulse wave velocity (PWV/PWA) will be performed at baseline and 2 hours following either a single dose oral antioxidant cocktail (1000 mg of Vitamin C, 600 IU of Vitamin E, and 600 mg of alpha-lipoic acid) or placebo on two days separated by at least 72 hours. Nitroglycerin mediated dilation (NMD, 0.4mg sub-lingual nitroglycerin spray), will be assessed at baseline.

Part two: Subjects, if interested will undergo a subcutaneous gluteal/hip fat biopsy. Micro vessels will be isolated from the adipose tissue and analyzed by pressurized myography for endothelial function and nitric oxide bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* documented childhood SES
* men and premenopausal women ages 18-40
* lean/overweight/or obese with BMI< or equal to 39kg/m2

Exclusion Criteria:

* cardiovascular, renal, pulmonary, hepatic, cerebral, or metabolic,disease
* use medications that affect vascular tone
* post menopausal women
* have class 3 obesity or BMI over 40

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-04; Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Acute Change in Flow mediated dilation | Change from baseline (2 hours)
  Flow-Mediated Dilation will be determined at baseline and 2 hours following acute antioxidant treatment

SECONDARY OUTCOMES:
Acute Change in Biomarkers of oxidative stress | Change from baseline (2 hours)
  Nitrite/nitrate, antioxidant capacity, and 8-isoprostane at baseline and 2 hours following acute antioxidant treatment
Acute Change in Arterial Stiffness | Change from baseline (2 hours)
  Pulse wave velocity will be determined at baseline and 2 hours following acute antioxidant treatment
Acute change in Flow mediated dilation | Immediate
  Nitroglycerin mediated dilation will be measured immediately following an administered 0.4mg dose of nitroglycerin spray, sub-lingual.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute , Georgia Regents University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes